CLINICAL TRIAL: NCT02931526
Title: Pharmacokinetics of Tigecycline in Critical Ill Patients Undergoing Continuous Renal Replacement Therapy
Brief Title: Study of Tigecycline Pharmacokinetics in Patients Undergoing Continuous Renal Replacement Therapy(CRRT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LCYJ1
Record Dates: First submitted 2016-09-19; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-07

CONDITIONS: Bacterial Infection; Critically Ill
Keywords: Tigecycline; Continuous Renal Replacement Therapy; Pharmacokinetics
MeSH Terms: conditions — Bacterial Infections; Critical Illness | interventions — Tigecycline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood, serum, urine, effluent fluid from dialysis machine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group CRRT: Patients who need to treat with tigecycline for bacterial infection, have renal insufficiency and have to treat with CRRT
  Interventions: Drug: Tigecycline
- Group non-CRRT: Patients who need to treat with tigecycline for bacterial infection, have normal renal function in ICU and have no need to treat with CRRT
  Interventions: Drug: Tigecycline

INTERVENTIONS:
Drug: Tigecycline — Patients who have the definitive diagnosis to treat with tigecycline for bacterial infection will be started on tigecycline with a loading dose 200mg IV followed by 100mg IV every 12h.
  Other Names: Tygacil

SUMMARY:
The aim of this study is to determine the Pharmacokinetics/Pharmacodynamics(PK/PD) of tigecycline in critical ill patients undergoing continuous renal replacement therapy（CRRT）and examine whether the dosage needs adjustment.

The study will observe two groups of patients respectively and compare the difference between them. Patients who need to receive CRRT when treat with high-dose tigecycline will be collected in Group CRRT. Patients who treat with high-dose tigecycline only will be collected in Group non-CRRT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years,hospitalized ICU patients, male or female;
* having definitive diagnosis to treat with tigecycline for bacterial infection;
* receiving CRRT with renal insufficiency or not receiving CRRT with normal renal function.

Exclusion Criteria:

* Patients with Child-Pugh C cirrhosis;
* Allergic to tetracycline or tigecycline;
* Patients received CRRT for < 3 days or treated with tigecycline < 3 days;
* Patients who are pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized Intensive Care Unit(ICU) patients in Zhujiang Hospital, in need of treatment with antiinfectives
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Tigecycline Steady State Plasma Concentrations | Day 1-3
  Steady State Plasma Concentration(Css) in blood

SECONDARY OUTCOMES:
Peak Plasma Concentration(Cmax) of Tigecycline in blood | Day 1-3
Trough Plasma Concentration(Cmin) of Tigecycline in blood | Day 1-3
Area Under the Plasma Concentration versus Time Curve(AUC) | Day 1-3
Minimal Inhibitory Concentration(MIC) | Day 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Wang Liqing, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhao HH, Tang WJ, Yang YX, Cen ZR, Wang LQ. PK/PD study of tigecycline in severely infected patients with continuous renal replacement therapy. Int J Clin Pharmacol Ther. 2020 Oct;58(10):531-538. doi: 10.5414/CP203669. PMID 32716292